CLINICAL TRIAL: NCT01779609
Title: Effect of a Dual ET(Endothelin)-Blocker on Exercise Induced Vascular Adaptations in Type 2 Diabetes Mellitus (T2DM)
Brief Title: ET-blockade and Exercise-induced Vascular Adaptations in T2DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ET-EX-TRAINING
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Bosentan; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bosentan + Exercise (Experimental): 2x/day 62.5 mg Bosentan for 4 weeks alongside 3x/week supervised exercise 2x/day 125 mg Bosentan for 4 weeks alongside 3x/week supervised exercise
  Interventions: Drug: Bosentan; Behavioral: Exercise
- Placebo + Exercise (Placebo Comparator): 2x/day 62.5 mg Placebo for 4 weeks alongside 3x/week supervised exercise 2x/day 125 mg Placebo for 4 weeks alongside 3x/week supervised exercise
  Interventions: Drug: Placebo; Behavioral: Exercise
- Exercise (Other): 3x/week supervised exercise for 8 weeks
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Drug: Bosentan
  Other Names: Tracleer; actelion pharmaceuticals
  Arms: Bosentan + Exercise
Drug: Placebo
  Other Names: actelion pharmaceuticals
  Arms: Placebo + Exercise
Behavioral: Exercise — Supervised exercise training program of 8 weeks, for 3x/week
  Other Names: Supervised Exercise Training Program

SUMMARY:
The purpose of this study is to establish the effect of ET blockade on vascular adaptations during an 8-week exercise program in subjects with T2DM. We hypothesize that combining ET - blockade with exercise training leads to an acute increase of exercise induced blood flow when compared with exercise alone. We expect that this will lead to an optimization of vascular training effect in T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus (>2 years since diagnosis) OR controls

Exclusion Criteria:

* <40 years of age
* >65 years of age
* smoking
* cardiovascular disease
* diabetes related manifest vascular complications
* Type 1 Diabetes Mellitus
* use of Glibenclamide
* use of HIV drugs
* use of calcineurin inhibitors
* use of drugs that interfere with CYP3A4 and CYP2C19

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Flow mediated dilation | 8 weeks

SECONDARY OUTCOMES:
Conduit Artery Dilator Capacity | 8 weeks
Intima-Media Thickness | 8 weeks
Maximal Oxygen Uptake | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Schreuder TH, Duncker DJ, Hopman MT, Thijssen DH. Randomized controlled trial using bosentan to enhance the impact of exercise training in subjects with type 2 diabetes mellitus. Exp Physiol. 2014 Nov;99(11):1538-47. doi: 10.1113/expphysiol.2014.081182. Epub 2014 Aug 28. PMID 25172889